CLINICAL TRIAL: NCT03767478
Title: Neuromuscular Electrical Stimulation For The Treatment Of Diabetic Neuropathy: A Multicentre, Double-blind, Pilot, Randomised, Sham-controlled Trial
Brief Title: Neuromuscular Electrical Stimulation For The Treatment of Diabetic Neuropathy
Acronym: NMES-DN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Actegy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18HH4610; IRAS ID (Other: 23712); NRES REC ID (Other: 18/NE/0281)
Record Dates: First submitted 2018-11-27; First posted 2018-12-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Peripheral Neuropathy; Diabetic Neuropathies; Diabetic Polyneuropathy; Diabetic Complication
Keywords: Neuromuscular electrical stimulation; Nerve conduction
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Complications

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Sham Comparator): Standard of Care + Sham Revitive Medic Coach (Sham Neuromuscular Electrical Stimulation Device) for 12 weeks
  Interventions: Device: Sham Revitive Medic Coach (Actegy Ltd)
- Intervention group (Active Comparator): Standard of Care + Revitive Medic Coach (Neuromuscular Electrical Stimulation Device) for 12 weeks
  Interventions: Device: Revitive Medic Coach (Actegy Ltd)

INTERVENTIONS:
Device: Revitive Medic Coach (Actegy Ltd) — Use the device for two 30-minute sessions per day, a minimum of five hours per week for 12 weeks at suprathreshold (2 x motor threshold).
  Other Names: Footplate Neuromuscular Electrical Stimulation Device
  Arms: Intervention group
Device: Sham Revitive Medic Coach (Actegy Ltd) — Use the device for two 30-minute sessions per day, a minimum of five hours per week for 12 weeks at suprathreshold (2 x motor threshold).
  Other Names: Sham Footplate Neuromuscular Electrical Stimulation Device
  Arms: Control group

SUMMARY:
Diabetic neuropathy (DN) is the most common complication of diabetes, affecting almost 50% of people with diabetes over the course of their lives. Symptoms vary from numbness to burning, aching and hypersensitivity in the lower limbs, indicative of sensory nerve loss. Motor neurons can also be affected, leading to muscle weakness and mobility issues, thus preventing patients from engaging in daily routines. Further sequelae include foot ulceration and Charcot neuroarthropathy, which are risk factors for lower limb amputation and mortality. In the United Kingdom, the annual costs of DN alone exceed £300 million, with further complications expected to cost an additional £1 billion. Currently, management strategies for DN focus on prevention and pain management. Neuromuscular electrical stimulation (NMES) is a novel nonpharmacological intervention for people with DN. NMES is the application of electrical impulses which are of sufficiency intensity to improve artificial contraction of the muscle tissue and may help with DN by improving nerve conductivity through direct stimulation of the nerves.

ELIGIBILITY:
INCLUSION CRITERIA

* Aged ≥18 (no upper limit)
* Diagnosis of type 1 or type 2 diabetes based on World Health Organisation (WHO) definition
* Diagnosis of diabetic neuropathy based on validated screening questionnaire Michigan Neuropathy Screening Instrument score of ≥4
* Access to internet at home to use the Revitive App (study smartphones will be provided)

EXCLUSION CRITERIA

* Lacks capacity to provide informed consent
* Pregnant
* Implanted electronic, cardiac or defibrillator device
* Other cause of peripheral neuropathy
* Current foot ulceration
* Severe vascular disease requiring invasive intervention
* Being treated for, or have the symptoms of, an existing deep vein thrombosis (DVT)
* Used a neuromuscular electrical stimulation (NMES) device within 1 year of randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure: neuropathy symptoms measured using validated screening questionnaire, Michigan Neuropathy Screening Instrument (MNSI) Part A questionnaire. | Week 6, Week 12, Week 26

SECONDARY OUTCOMES:
Feasibility outcome measure: recruitment rate measured using screening and randomisation logs. | Pre-screening / Identification, Recruitment and Consent, Baseline
Feasibility outcome measure: participant retention rate measured using randomisation and withdrawal logs. | Recruitment and Consent, Baseline, Week 12, Week 26
Feasibility outcome measure: adherence to treatment measured using Revitive App and a patient diary. | Week 12
Safety outcome measure: Adverse Events (AEs) collected and reported via AE form. | Baseline, Week 3, Week 6, Week 9, Week 12, Week 26 (and any communication in between)
Safety outcome measure: Adverse Device Effects (ADEs) collected and reported via AE form. | Baseline, Week 3, Week 6, Week 9, Week 12, Week 26 (and any communication in between)
Safety outcome measure: Serious Adverse Events (SAEs) collected and reported via SAE form. | Baseline, Week 3, Week 6, Week 9, Week 12, Week 26 (and any communication in between)
Safety outcome measure: Serious Adverse Device Effects (SADEs) collected and reported via SAE form. | Baseline, Week 3, Week 6, Week 9, Week 12, Week 26 (and any communication in between)
Secondary outcome measure: sural nerve conductivity measured using a nerve conduction study (central site only). | Week 12, Week 26.
  Nerve conduction parameters include sural nerve conduction velocity (m/s) and SNAP amplitude (µV).
Secondary outcome measure: superficial peroneal nerve conductivity measured using a nerve conduction study (central site only). | Week 12, Week 26
  Nerve conduction parameters include conduction velocity (m/s), calculated using distance and latency (ms), and SNAP amplitude (μV).
Secondary outcome measure: common peroneal nerve conductivity measured using a nerve conduction study (central site only). | Week 12, Week 26
  Nerve conduction parameters include conduction velocity (m/s), calculated using distance and distal latency (ms), Compound Muscle Action Potential (CMAP) amplitude (mV) and minimum F wave latency (ms).
Secondary outcome measure: tibial nerve conductivity measured using a nerve conduction study (central site only). | Week 12, Week 26
  Nerve conduction parameters include conduction velocity (m/s), calculated using distance and distal latency (ms), Compound Muscle Action Potential (CMAP) amplitude (mV) and minimum F wave latency (ms).
Secondary outcome measure: somatosensory nerve fibre function measured using QuantitativeSensory Testing (QST) (central site only). | Week 12, Week 26
  Somatosensory nerve fibre function will be assessed using the German Research Network on Neuropathic Pain (DFNS) QST protocol. The battery of tests includes measures of cold and warm detection thresholds, paradoxical heat sensations, cold and heat pain thresholds, mechanical detection threshold, mechanical pain threshold, mechanical pain sensitivity, dynamic mechanical allodynia, temporal pain summation, vibration detection threshold and pressure pain threshold.
Secondary outcome measure: blood glucose measured using HbA1c. | Week 12
Secondary outcome measure: mobility and balance measured using validated Berg Balance Scale (BBS). | Week 12, Week 26
Secondary outcome measure: neuropathy signs measured using validated screening questionnaire, Michigan Neuropathy Screening Instrument (MNSI) Part B questionnaire. | Week 12, Week 26
Secondary outcome measure: symptoms measured using Total Symptom Score (TSS). | Week 12
Secondary outcome measure: protected sensation measured using monofilament test. | Week 12, Week 26
Secondary outcome measure: neuropathic pain measured using Neuropathic Pain Symptom Inventory (NPSI). | Week 12, Week 26
Secondary outcome measure: device sensation measured using device sensory threshold and suprathreshold. | Week 12, Week 26
Secondary outcome measure: device experience measured using device experience questionnaire. | Week 12
Secondary outcome measure: device credibility and expectancy measured using modified credibility and expectancy questionnaire. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alun H Davies, MA DM DSC FRCS FEBVS, Study Chair — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Available on request.
Supporting Information: Study Protocol, SAP

DOCUMENTS (1):
  • Study Protocol (2025-01-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT03767478/Prot_000.pdf